CLINICAL TRIAL: NCT04027049
Title: Biologic Mechanisms of Early Exercise After Intracerebral Hemorrhage: a Pilot Randomized Controlled Trial of Cycle Ergometry
Brief Title: Biologic Mechanisms of Early Exercise After Intracerebral Hemorrhage
Acronym: BEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00154440
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Intracerebral Hemorrhage; Acute Ischemic Stroke
Keywords: rehabilitation; cycle ergometry
MeSH Terms: conditions — Cerebral Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Pilot randomized parallel group design
Who Masked: Outcomes Assessor
Masking Description: The clinician assessing outcomes will not have been involved in the care of the patient and will not be aware of the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Supine cycle ergometry of the lower extremities (Experimental): Patients will receive two 20 minute cycle ergometry sessions separated by at least 4 hours in addition to usual care. The cycle will be set to a gear of zero and will begin in passive mode, the patient will be able to actively cycle if patients are able.
  Interventions: Device: Supine cycle ergometry of the lower extremities
- Control (No Intervention): Patients will receive usual care only.

INTERVENTIONS:
Device: Supine cycle ergometry of the lower extremities — The cycle ergometer allows for movement of the lower extremities by a motor if a patient is experiencing a disorder of consciousness or is otherwise unable to move one or both legs. If a patient is able to cycle actively the device allows the patient to move patient's legs without support of the motor.
  Arms: Supine cycle ergometry of the lower extremities

SUMMARY:
This study aims to determine whether in-bed cycle ergometry, early in the hospital course after a brain hemorrhage could balance damaging and reparative inflammation in the brain. Inflammatory factors of two groups of patients with brain hemorrhage will be compared, one group will receive in-bed cycling beginning 3 days after hemorrhage plus usual care and the other group will receive usual care only.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial intracerebral hemorrhage with or without intraventricular hemorrhage
* Pre-morbid modified Rankin Score of 0-2
* Patient must be able to provide informed consent or have a legally authorized representative to provide consent on patient's behalf

Exclusion Criteria:

* Patients with known inflammatory conditions, infection requiring antibiotics or pregnancy
* Patients receiving daily anti-inflammatory medications including but not limited to prednisone, methotrexate, non-steroidal anti-inflammatory medications (ibuprofen, naproxen, indomethacin, celecoxib) and aspirin >325mg
* Glasgow Coma Score (GCS) 3 48 hours after admission
* Patients in whom withdrawal of life support is being considered by surrogate decision makers
* Injury to the lower extremities, hips or pelvis, weight >250 kg (weight limit of cycle), or body habitus precluding normal function of cycle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Zink, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Department of Neurology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amidei C, Sole ML. Physiological responses to passive exercise in adults receiving mechanical ventilation. Am J Crit Care. 2013 Jul;22(4):337-48. doi: 10.4037/ajcc2013284. PMID 23817823
- [Background] Arafah BM, Nishiyama FJ, Tlaygeh H, Hejal R. Measurement of salivary cortisol concentration in the assessment of adrenal function in critically ill subjects: a surrogate marker of the circulating free cortisol. J Clin Endocrinol Metab. 2007 Aug;92(8):2965-71. doi: 10.1210/jc.2007-0181. Epub 2007 May 29. PMID 17535998
- [Background] Burn JP. Reliability of the modified Rankin Scale. Stroke. 1992 Mar;23(3):438. No abstract available. PMID 1610453
- [Background] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Background] Calabrese EJ. Pre- and post-conditioning hormesis in elderly mice, rats, and humans: its loss and restoration. Biogerontology. 2016 Aug;17(4):681-702. doi: 10.1007/s10522-016-9646-8. Epub 2016 Apr 13. PMID 27075594
- [Background] Camargo Pires-Neto R, Fogaca Kawaguchi YM, Sayuri Hirota A, Fu C, Tanaka C, Caruso P, Park M, Ribeiro Carvalho CR. Very early passive cycling exercise in mechanically ventilated critically ill patients: physiological and safety aspects--a case series. PLoS One. 2013 Sep 9;8(9):e74182. doi: 10.1371/journal.pone.0074182. eCollection 2013. PMID 24040200
- [Background] Chen J, Qin J, Su Q, Liu Z, Yang J. Treadmill rehabilitation treatment enhanced BDNF-TrkB but not NGF-TrkA signaling in a mouse intracerebral hemorrhage model. Neurosci Lett. 2012 Oct 31;529(1):28-32. doi: 10.1016/j.neulet.2012.09.021. Epub 2012 Sep 19. PMID 22999926
- [Background] Cocks K, Torgerson DJ. Sample size calculations for pilot randomized trials: a confidence interval approach. J Clin Epidemiol. 2013 Feb;66(2):197-201. doi: 10.1016/j.jclinepi.2012.09.002. Epub 2012 Nov 27. PMID 23195919
- [Background] Di Napoli M, Godoy DA, Campi V, Masotti L, Smith CJ, Parry Jones AR, Hopkins SJ, Slevin M, Papa F, Mogoanta L, Pirici D, Popa Wagner A. C-reactive protein in intracerebral hemorrhage: time course, tissue localization, and prognosis. Neurology. 2012 Aug 14;79(7):690-9. doi: 10.1212/WNL.0b013e318264e3be. Epub 2012 Aug 1. PMID 22855859
- [Background] Duffy L, Gajree S, Langhorne P, Stott DJ, Quinn TJ. Reliability (inter-rater agreement) of the Barthel Index for assessment of stroke survivors: systematic review and meta-analysis. Stroke. 2013 Feb;44(2):462-8. doi: 10.1161/STROKEAHA.112.678615. Epub 2013 Jan 8. PMID 23299497
- [Background] Fearon P, McArthur KS, Garrity K, Graham LJ, McGroarty G, Vincent S, Quinn TJ. Prestroke modified rankin stroke scale has moderate interobserver reliability and validity in an acute stroke setting. Stroke. 2012 Dec;43(12):3184-8. doi: 10.1161/STROKEAHA.112.670422. Epub 2012 Nov 13. PMID 23150650
- [Background] Fogelholm R, Murros K, Rissanen A, Avikainen S. Long term survival after primary intracerebral haemorrhage: a retrospective population based study. J Neurol Neurosurg Psychiatry. 2005 Nov;76(11):1534-8. doi: 10.1136/jnnp.2004.055145. PMID 16227546
- [Background] Gao Z, Wang J, Thiex R, Rogove AD, Heppner FL, Tsirka SE. Microglial activation and intracerebral hemorrhage. Acta Neurochir Suppl. 2008;105:51-3. doi: 10.1007/978-3-211-09469-3_11. PMID 19066082
- [Background] Giraldo E, Garcia JJ, Hinchado MD, Ortega E. Exercise intensity-dependent changes in the inflammatory response in sedentary women: role of neuroendocrine parameters in the neutrophil phagocytic process and the pro-/anti-inflammatory cytokine balance. Neuroimmunomodulation. 2009;16(4):237-44. doi: 10.1159/000212384. Epub 2009 Apr 9. PMID 19365147
- [Background] Gomez-Cabrera MC, Domenech E, Vina J. Moderate exercise is an antioxidant: upregulation of antioxidant genes by training. Free Radic Biol Med. 2008 Jan 15;44(2):126-31. doi: 10.1016/j.freeradbiomed.2007.02.001. Epub 2007 Feb 9. PMID 18191748
- [Background] Guo YC, Song XK, Xu YF, Ma JB, Zhang JJ, Han PJ. The expression and mechanism of BDNF and NGB in perihematomal tissue in rats with intracerebral hemorrhage. Eur Rev Med Pharmacol Sci. 2017 Aug;21(15):3452-3458. PMID 28829495
- [Background] Hanley DF. Intraventricular hemorrhage: severity factor and treatment target in spontaneous intracerebral hemorrhage. Stroke. 2009 Apr;40(4):1533-8. doi: 10.1161/STROKEAHA.108.535419. Epub 2009 Feb 26. PMID 19246695
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Hemphill JC 3rd, Farrant M, Neill TA Jr. Prospective validation of the ICH Score for 12-month functional outcome. Neurology. 2009 Oct 6;73(14):1088-94. doi: 10.1212/WNL.0b013e3181b8b332. Epub 2009 Sep 2. PMID 19726752
- [Background] Hermans G, Clerckx B, Vanhullebusch T, Segers J, Vanpee G, Robbeets C, Casaer MP, Wouters P, Gosselink R, Van Den Berghe G. Interobserver agreement of Medical Research Council sum-score and handgrip strength in the intensive care unit. Muscle Nerve. 2012 Jan;45(1):18-25. doi: 10.1002/mus.22219. PMID 22190301
- [Background] Hodgson CL, Stiller K, Needham DM, Tipping CJ, Harrold M, Baldwin CE, Bradley S, Berney S, Caruana LR, Elliott D, Green M, Haines K, Higgins AM, Kaukonen KM, Leditschke IA, Nickels MR, Paratz J, Patman S, Skinner EH, Young PJ, Zanni JM, Denehy L, Webb SA. Expert consensus and recommendations on safety criteria for active mobilization of mechanically ventilated critically ill adults. Crit Care. 2014 Dec 4;18(6):658. doi: 10.1186/s13054-014-0658-y. PMID 25475522
- [Background] Ishida A, Misumi S, Ueda Y, Shimizu Y, Cha-Gyun J, Tamakoshi K, Ishida K, Hida H. Early constraint-induced movement therapy promotes functional recovery and neuronal plasticity in a subcortical hemorrhage model rat. Behav Brain Res. 2015 May 1;284:158-66. doi: 10.1016/j.bbr.2015.02.022. Epub 2015 Feb 17. PMID 25700666
- [Background] Ji LL, Gomez-Cabrera MC, Vina J. Exercise and hormesis: activation of cellular antioxidant signaling pathway. Ann N Y Acad Sci. 2006 May;1067:425-35. doi: 10.1196/annals.1354.061. PMID 16804022
- [Background] Kimawi I, Lamberjack B, Nelliot A, Toonstra AL, Zanni J, Huang M, Mantheiy E, Kho ME, Needham DM. Safety and Feasibility of a Protocolized Approach to In-Bed Cycling Exercise in the Intensive Care Unit: Quality Improvement Project. Phys Ther. 2017 Jun 1;97(6):593-602. doi: 10.1093/ptj/pzx034. PMID 28379571
- [Background] Kho ME, Martin RA, Toonstra AL, Zanni JM, Mantheiy EC, Nelliot A, Needham DM. Feasibility and safety of in-bed cycling for physical rehabilitation in the intensive care unit. J Crit Care. 2015 Dec;30(6):1419.e1-5. doi: 10.1016/j.jcrc.2015.07.025. Epub 2015 Jul 29. PMID 26318234
- [Background] Kho ME, Molloy AJ, Clarke FJ, Ajami D, McCaughan M, Obrovac K, Murphy C, Camposilvan L, Herridge MS, Koo KK, Rudkowski J, Seely AJ, Zanni JM, Mourtzakis M, Piraino T, Cook DJ; Canadian Critical Care Trials Group. TryCYCLE: A Prospective Study of the Safety and Feasibility of Early In-Bed Cycling in Mechanically Ventilated Patients. PLoS One. 2016 Dec 28;11(12):e0167561. doi: 10.1371/journal.pone.0167561. eCollection 2016. PMID 28030555
- [Background] Lei C, Lin S, Zhang C, Tao W, Dong W, Hao Z, Liu M, Wu B. High-mobility group box1 protein promotes neuroinflammation after intracerebral hemorrhage in rats. Neuroscience. 2013 Jan 3;228:190-9. doi: 10.1016/j.neuroscience.2012.10.023. Epub 2012 Oct 22. PMID 23085216
- [Background] Mello RC, Sad EF, Andrade BC, Neves SP, Santos SM, Sarquis MM, Marik PE, Dias EP. Serum and salivary cortisol in the diagnosis of adrenal insufficiency and as a predictor of the outcome in patients with severe sepsis. Arq Bras Endocrinol Metabol. 2011 Oct;55(7):455-9. doi: 10.1590/s0004-27302011000700004. PMID 22147093
- [Background] Mendelow AD, Gregson BA, Rowan EN, Murray GD, Gholkar A, Mitchell PM; STICH II Investigators. Early surgery versus initial conservative treatment in patients with spontaneous supratentorial lobar intracerebral haematomas (STICH II): a randomised trial. Lancet. 2013 Aug 3;382(9890):397-408. doi: 10.1016/S0140-6736(13)60986-1. Epub 2013 May 29. PMID 23726393
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Ortega E. The
- [Background] Ovbiagele B, Goldstein LB, Higashida RT, Howard VJ, Johnston SC, Khavjou OA, Lackland DT, Lichtman JH, Mohl S, Sacco RL, Saver JL, Trogdon JG; American Heart Association Advocacy Coordinating Committee and Stroke Council. Forecasting the future of stroke in the United States: a policy statement from the American Heart Association and American Stroke Association. Stroke. 2013 Aug;44(8):2361-75. doi: 10.1161/STR.0b013e31829734f2. Epub 2013 May 22. PMID 23697546
- [Background] Poon MT, Fonville AF, Al-Shahi Salman R. Long-term prognosis after intracerebral haemorrhage: systematic review and meta-analysis. J Neurol Neurosurg Psychiatry. 2014 Jun;85(6):660-7. doi: 10.1136/jnnp-2013-306476. Epub 2013 Nov 21. PMID 24262916
- [Background] Quinn TJ, Dawson J, Walters MR, Lees KR. Reliability of the modified Rankin Scale: a systematic review. Stroke. 2009 Oct;40(10):3393-5. doi: 10.1161/STROKEAHA.109.557256. Epub 2009 Aug 13. PMID 19679846
- [Background] Qureshi AI, Palesch YY, Barsan WG, Hanley DF, Hsu CY, Martin RL, Moy CS, Silbergleit R, Steiner T, Suarez JI, Toyoda K, Wang Y, Yamamoto H, Yoon BW; ATACH-2 Trial Investigators and the Neurological Emergency Treatment Trials Network. Intensive Blood-Pressure Lowering in Patients with Acute Cerebral Hemorrhage. N Engl J Med. 2016 Sep 15;375(11):1033-43. doi: 10.1056/NEJMoa1603460. Epub 2016 Jun 8. PMID 27276234
- [Background] Steins Bisschop CN, Courneya KS, Velthuis MJ, Monninkhof EM, Jones LW, Friedenreich C, van der Wall E, Peeters PH, May AM. Control group design, contamination and drop-out in exercise oncology trials: a systematic review. PLoS One. 2015 Mar 27;10(3):e0120996. doi: 10.1371/journal.pone.0120996. eCollection 2015. PMID 25815479
- [Background] Takamatsu Y, Tamakoshi K, Waseda Y, Ishida K. Running exercise enhances motor functional recovery with inhibition of dendritic regression in the motor cortex after collagenase-induced intracerebral hemorrhage in rats. Behav Brain Res. 2016 Mar 1;300:56-64. doi: 10.1016/j.bbr.2015.12.003. Epub 2015 Dec 7. PMID 26675889
- [Background] Franca EE, Ribeiro LC, Lamenha GG, Magalhaes IK, Figueiredo TG, Costa MJ, Elihimas UF Junior, Feitosa BL, Andrade MD, Correia MA Junior, Ramos FF, Castro CM. Oxidative stress and immune system analysis after cycle ergometer use in critical patients. Clinics (Sao Paulo). 2017 Mar;72(3):143-149. doi: 10.6061/clinics/2017(03)03. PMID 28355359
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Thelandersson A, Nellgard B, Ricksten SE, Cider A. Effects of Early Bedside Cycle Exercise on Intracranial Pressure and Systemic Hemodynamics in Critically Ill Patients in a Neurointensive Care Unit. Neurocrit Care. 2016 Dec;25(3):434-439. doi: 10.1007/s12028-016-0278-2. PMID 27216931
- [Background] Wang P, Li CG, Qi Z, Cui D, Ding S. Acute exercise stress promotes Ref1/Nrf2 signalling and increases mitochondrial antioxidant activity in skeletal muscle. Exp Physiol. 2016 Mar;101(3):410-20. doi: 10.1113/EP085493. Epub 2016 Jan 23. PMID 26682532
- [Background] Wang XM, Zhang YG, Li AL, Long ZH, Wang D, Li XX, Xia JH, Luo SY, Shan YH. Expressions of serum inflammatory cytokines and their relationship with cerebral edema in patients with acute basal ganglia hemorrhage. Eur Rev Med Pharmacol Sci. 2016 Jul;20(13):2868-71. PMID 27424987
- [Background] Wei P, You C, Jin H, Chen H, Lin B. Correlation between serum IL-1beta levels and cerebral edema extent in a hypertensive intracerebral hemorrhage rat model. Neurol Res. 2014 Feb;36(2):170-5. doi: 10.1179/1743132813Y.0000000292. Epub 2013 Dec 19. PMID 24410061
- [Background] Winkelman C. Investigating activity in hospitalized patients with chronic obstructive pulmonary disease: a pilot study. Heart Lung. 2010 Jul-Aug;39(4):319-30. doi: 10.1016/j.hrtlng.2009.09.004. Epub 2010 Apr 8. PMID 20561844
- [Background] Wu J, Yang S, Xi G, Song S, Fu G, Keep RF, Hua Y. Microglial activation and brain injury after intracerebral hemorrhage. Acta Neurochir Suppl. 2008;105:59-65. doi: 10.1007/978-3-211-09469-3_13. PMID 19066084
- [Background] Xue M, Del Bigio MR. Comparison of brain cell death and inflammatory reaction in three models of intracerebral hemorrhage in adult rats. J Stroke Cerebrovasc Dis. 2003 May-Jun;12(3):152-9. doi: 10.1016/S1052-3057(03)00036-3. PMID 17903920
- [Background] Yang X, Ren W, Zu H, Dong Q. Evaluate the serum cortisol in patients with intracerebral hemorrhage. Clin Neurol Neurosurg. 2014 Aug;123:127-30. doi: 10.1016/j.clineuro.2014.05.019. Epub 2014 Jun 5. PMID 25012024
- [Background] Yang Z, Yu A, Liu Y, Shen H, Lin C, Lin L, Wang S, Yuan B. Regulatory T cells inhibit microglia activation and protect against inflammatory injury in intracerebral hemorrhage. Int Immunopharmacol. 2014 Oct;22(2):522-5. doi: 10.1016/j.intimp.2014.06.037. Epub 2014 Jul 4. PMID 25000335
- [Background] Yong MS, Hwangbo K. Skilled reach training influences brain recovery following intracerebral hemorrhage in rats. J Phys Ther Sci. 2014 Mar;26(3):405-7. doi: 10.1589/jpts.26.405. Epub 2014 Mar 25. PMID 24707093
- [Background] Yuan ZH, Jiang JK, Huang WD, Pan J, Zhu JY, Wang JZ. A meta-analysis of the efficacy and safety of recombinant activated factor VII for patients with acute intracerebral hemorrhage without hemophilia. J Clin Neurosci. 2010 Jun;17(6):685-93. doi: 10.1016/j.jocn.2009.11.020. PMID 20399668
- [Background] Zhao X, Sun G, Ting SM, Song S, Zhang J, Edwards NJ, Aronowski J. Cleaning up after ICH: the role of Nrf2 in modulating microglia function and hematoma clearance. J Neurochem. 2015 Apr;133(1):144-52. doi: 10.1111/jnc.12974. Epub 2014 Nov 24. PMID 25328080

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Started | 14 | 11
Completed | 12 | 11
Not Completed | 2 | 0
Not completed — Withdrawn by family | 1 | 0
Not completed — Participant safety | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (14.3) | 62.3 (18.4) | 65.8 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 11 | 25
Type of Stroke [Count of Participants; unit: Participants]
  Acute Ischemic | 5 | 4 | 9
  Intracerebral Hemorrhage | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Interleukin-1beta Level in Blood (Picogram/Milliliter)
Time Frame: Day 1, day 3 and day 7 of study
Population: Samples collected did not meet the threshold for analysis, therefore this outcome measure could not be assessed.
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Absolute Change in Interleukin-6 Level in Blood (Picogram/Milliliter)
Time Frame: Day 1, day 3 and day 7 of study
Population: One participant was withdrawn for safety reasons in the intervention arm. All timepoints collected are reported.
Measure: Median (Inter-Quartile Range); unit: picogram/milliliter
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 13 | 11
picogram/milliliter
  Day 1 | 7.01 [1.89 to 10.51] | 6.18 [2.27 to 15.68]
  Day 3: number analyzed (Participants) | 11 | 11
  Day 3 | 4.3 [1.89 to 10.94] | 4.59 [2.26 to 9.12]
  Day 7: number analyzed (Participants) | 10 | 10
  Day 7 | 2.94 [1.91 to 12.36] | 3.17 [0.88 to 4.29]

3. Primary Outcome: Change in Tumor Necrosis Factor-alpha Level in Blood (Picogram/Milliliter)
Time Frame: Day 1, day 3 and day 7 of study
Population: Samples collected did not meet the threshold for analysis, therefore this outcome measure could not be assessed.
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in C Reactive Protein Level in Blood (Nanogram/Milliliter)
Time Frame: Day 1, day 3 and day 7 of study
Population: C reactive protein was not performed due to lack of funding.
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Absolute Change in Brain Derived Neurotrophic Factor Level in Blood (Picogram/Milliliter)
Time Frame: Day 1, day 3 and day 7 of study
Population: Participants who were able to have samples drawn are reported.
Measure: Median (Inter-Quartile Range); unit: picograms/mL
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 13 | 11
picograms/mL
  Day 1 | 8038.53 [2980.91 to 11669.31] | 2554.34 [1945.37 to 4223.35]
  Day 3: number analyzed (Participants) | 11 | 11
  Day 3 | 4380.57 [3706.41 to 7369.67] | 3043.86 [1204.4 to 4536.79]
  Day 7: number analyzed (Participants) | 10 | 10
  Day 7 | 3979.26 [2274.52 to 6745.13] | 2494.29 [1012.11 to 2812.83]

6. Primary Outcome: Change in Interleukin-1beta Level in Cerebrospinal Fluid (Picogram/Milliliter)
Description: Cerebrospinal fluid (CSF) will be collected only in patients with an external ventricular drain as part of patients' care.
Time Frame: Day 1, day 3 and day 7 of study
Population: Samples collected did not meet the threshold for analysis, therefore this outcome measure could not be assessed.
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Absolute Change in Interleukin-6 Level in CSF (Picogram/Milliliter)
Description: CSF will be collected only in patients with an external ventricular drain as part of patients' care.
Time Frame: Day 1, day 3 and day 7 of study
Population: 4 participants had an external ventricular drain and had CSF collected (2 intervention, 2 control)
Measure: Number; unit: picograms/mL
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 2 | 2
picograms/mL
  First participant in each arm, day 1: number analyzed (Participants) | 1 | 1
  First participant in each arm, day 1 | 1659 | 158.79
  First participant in each arm, day 3: number analyzed (Participants) | 1 | 1
  First participant in each arm, day 3 | 3379.57 | 386.02
  First participant in each arm, day 7: number analyzed (Participants) | 1 | 1
  First participant in each arm, day 7 | 2729.16 | 19.2
  Second participant in each arm, day 1: number analyzed (Participants) | 1 | 1
  Second participant in each arm, day 1 | 268 | 454.64
  Second participant in each arm, day 3: number analyzed (Participants) | 1 | 1
  Second participant in each arm, day 3 | 495.57 | 1040.6
  Second participant in each arm, day 7: number analyzed (Participants) | 1 | 1
  Second participant in each arm, day 7 | 750.79 | 401.51

8. Primary Outcome: Change in Tumor Necrosis Factor (TNF) -Alpha Level in CSF (Picogram/Milliliter)
Description: CSF will be collected only in patients with an external ventricular drain as part of patients' care. TNF-alpha normal range (1.45 pg/mL to 1073.41 pg/mL)
Time Frame: Day 1, day 3 and day 7 of study
Population: Samples collected did not meet the threshold for analysis, therefore this outcome measure could not be assessed.
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Change in C Reactive Protein Level in CSF (Nanogram/Milliliter)
Description: CSF will be collected only in patients with an external ventricular drain as part of patients' care
Time Frame: Day 1, day 3 and day 7 of study
Population: C Reactive Protein assay was not performed due to lack of funding.
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Absolute Change in Brain Derived Neurotrophic Factor Level in CSF (Picogram/Milliliter)
Description: CSF will be collected only in patients with an external ventricular drain as part of patients' care
Time Frame: Day 1, day 3 and day 7 of study
Population: 4 participants had an external ventricular drain and had CSF collected (2 intervention, 2 control)
Measure: Number; unit: picograms/mL
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 2 | 2
picograms/mL
  First participant in each arm, day 1: number analyzed (Participants) | 1 | 1
  First participant in each arm, day 1 | 26.26 | 3.71
  First participant in each arm, day 3: number analyzed (Participants) | 1 | 1
  First participant in each arm, day 3 | 12.42 | 2.64
  First participant in each arm, day 7: number analyzed (Participants) | 1 | 1
  First participant in each arm, day 7 | 4.38 | 2.75
  Second participant in each arm, day 1: number analyzed (Participants) | 1 | 1
  Second participant in each arm, day 1 | 23.98 | 2.02
  Second participant in each arm, day 3: number analyzed (Participants) | 1 | 1
  Second participant in each arm, day 3 | 7.81 | 2.64
  Second participant in each arm, day 7: number analyzed (Participants) | 1 | 1
  Second participant in each arm, day 7 | 3.21 | 2.02

11. Primary Outcome: Change in Salivary Cortisol Level (Microgram/Deciliter)
Time Frame: Day 1, day 3 and day 7 of study
Population: Samples not collected
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Absolute Change in Hand-held Dynamometry Score (Pounds)
Description: An average of three hand-held dynamometry measurements will be calculated for each measurement episode and the change over time will be measured. Grip strength is reported in pounds and compared against population and sex-based normative values.
Time Frame: Study days 1, 3, 7, day of transfer from the ICU or discharge, whichever comes first, assessed up to 60 days
Population: Six participants, 3 in each group had dynamometry values collected.
Measure: Number; unit: pounds
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 3 | 3
pounds
  First participant in each arm, day 1: number analyzed (Participants) | 1 | 1
  First participant in each arm, day 1 | 28.8 | 25.7
  First participant in each arm, day 3: number analyzed (Participants) | 1 | 1
  First participant in each arm, day 3 | 19.87 | 24.55
  First participant in each arm, day 7: number analyzed (Participants) | 1 | 1
  First participant in each arm, day 7 | 21.2 | 33.6
  First participant in each arm, discharge: number analyzed (Participants) | 1 | 1
  First participant in each arm, discharge | 14.7 | 55.4
  Second participant in each arm, day 1: number analyzed (Participants) | 1 | 1
  Second participant in each arm, day 1 | 41.6 | 19.57
  Second participant in each arm, day 3: number analyzed (Participants) | 1 | 1
  Second participant in each arm, day 3 | 40.87 | 22.63
  Second participant in each arm, day 7: number analyzed (Participants) | 1 | 1
  Second participant in each arm, day 7 | 60.07 | 20.07
  Second participant in each arm, discharge: number analyzed (Participants) | 1 | 1
  Second participant in each arm, discharge | 48.33 | 10
  Third participant in each arm, day 1: number analyzed (Participants) | 1 | 1
  Third participant in each arm, day 1 | 91.5 | 70.97
  Third participant in each arm, day 3: number analyzed (Participants) | 1 | 1
  Third participant in each arm, day 3 | 92.9 | 87.53
  Third participant in each arm, day 7: number analyzed (Participants) | 1 | 1
  Third participant in each arm, day 7 | 79.4 | 75.76
  Third participant in each arm, discharge: number analyzed (Participants) | 1 | 1
  Third participant in each arm, discharge | 90.93 | 70.6

13. Secondary Outcome: Global Pre-morbid Physical Health Status as Measured by the Promis Scale v1.2
Description: The global physical health status subscale of the Promis scale v1.2 will be used to measure pre-morbid physical health status. A 5-point Likert scale is used to score each of the four items. The scores for each item are summed as a raw score and are converted to T scores using a standardized table with higher T scores indicating better physical health status. An average t score representing the population is 50. 10 points is equal to 1 standard deviation, thus a score of 60 means that one is one standard deviation better than the general population.
Time Frame: Day 1 of study
Population: Participants who completed the survey are reported.
Measure: Mean (Inter-Quartile Range); unit: T-score
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 6 | 5
T-score | 38.6 [37.4 to 43.63] | 44.9 [37.4 to 57.7]

14. Secondary Outcome: Global Pre-morbid Mental Health Status as Measured by the Promis Scale v1.2
Description: The global mental health status subscale of the Promis scale will be used to measure pre-morbid mental health status. A 5-point Likert scale is used to score each of the four items. The scores for each item are summed as a raw score and are converted to T scores using a standardized table with higher T scores indicating better physical health status. An average t score representing the population is 50. Ten points is equal to 1 standard deviation, thus a score of 60 means that one is one standard deviation better than the general population.
Time Frame: Day 1 of study
Population: Participants who completed the survey are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 6 | 6
score on a scale | 53.3 [45.95 to 53.3] | 41.15 [35.05 to 47.1]

15. Secondary Outcome: Functional Status as Assessed by the Modified Rankin Score (mRS)
Description: The modified Rankin score will be used to measure function in terms of activities of daily living after stroke. A six-point ordinal scale (0-6) with lower scores indicating less disability and higher scores indicating increasingly severe disability. A score of 6 indicates death. Reporting the frequency of each score category.
Time Frame: Standard of care 90-day assessment
Population: 17 patients had the modified Rankin assessed per standard of care at 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 7 | 10
Participants
  mRS 0 | 0 | 0
  mRS 1 | 2 | 0
  mRS 2 | 1 | 3
  mRS 3 | 0 | 1
  mRS 4 | 1 | 1
  mRS 5 | 2 | 2
  mRS 6 | 1 | 3

16. Secondary Outcome: Change in the Functional Status as Assessed by the Modified Rankin Score
Description: The modified Rankin score will be used to measure function in terms of activities of daily living after stroke. A six-point ordinal scale (0-6) with lower scores indicating less disability and higher scores indicating increasingly severe disability. A score of 6 indicates death. Change in functional status was calculated by subtracting the first score (discharge) from the second score (90 day assessment).
Time Frame: Day of ICU transfer or discharge, 90 day assessment
Population: Only 4 patients had scores at discharge or transfer and at the 90 day assessment per standard of care (1 in the treatment group and 3 in the control group). Change in scores are reported.
Measure: Number; unit: score on a scale
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 1 | 3
score on a scale
  First participant, change in score: number analyzed (Participants) | 1 | 1
  First participant, change in score | 0 | 2
  Second participant, change in score: number analyzed (Participants) | 0 | 1
  Second participant, change in score |  | -1
  Third participant, change in score: number analyzed (Participants) | 0 | 1
  Third participant, change in score |  | 2

17. Secondary Outcome: Change in Muscle Strength as Assessed by the Medical Research Council Sum (MRCS) Score
Description: The MRCS will be used to measure muscle strength over time. The instrument is a 60 point scale indicating muscle strength in 6 muscle groups. Three muscle groups each on the right and left upper extremities and three each in the right and left lower extremities. Each muscle group is scored from 0-5 out of a possible 5 points. A composite score with a maximum of 60 is produced, 30 points can be achieved for each side of the body.
Time Frame: Study days 1, 3, 7, On transfer from the ICU or discharge from the hospital, whichever comes first, assessed up to 60 days, 30-day follow-up visit
Population: Resource limitations precluded collection of this data.
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Ability to Perform Activities of Daily Living as Assessed by the Barthel Index
Description: The Barthel index will be used to measure a participant's ability to perform activities of daily living in detail. The instrument is a 10-item scale with a range of 0 -100 points. Higher scores indicate higher levels of function.
Time Frame: On transfer from the ICU or discharge from the hospital, whichever comes first, assessed up to 60 days, 30-day follow-up visit
Population: Due to resource constraints this assessment was only performed at discharge and only in 14 patients, 7 each in the intervention and control arms.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 7 | 7
score on a scale | 10 [2.5 to 25] | 5 [2.5 to 22.5]

19. Secondary Outcome: Health Status as Assessed by the Stroke Impact Scale Version 3.0
Description: This is a 59-item questionnaire that will measure health status in 8 domains following the stroke. A 5-point Likert scale is used to score each item with higher scores indicating higher perceived health status.
Time Frame: During the 30-day follow up visit
Population: Resource constraints precluded collection of this data.
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Perception of Stroke Recovery as Assessed by the Stroke Impact Scale Version 3.0
Description: The last question of the instrument measures a participant's perception of stroke recovery using a 0-100 scale with higher scores representing higher levels of recovery and lower scores representing less recovery.
Time Frame: During the 30-day follow up visit
Population: Resource constraints precluded collection of this data.
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 90 days
Arm/Group | Supine Cycle Ergometry of the Lower Extremities | Control
All-Cause Mortality (participants affected / at risk) | 1/14 | 3/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 2/14 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supine Cycle Ergometry of the Lower Extremities (N=14) | Control (N=11)
systolic blood pressure above goal (Cardiac disorders) | 1 (1) | 0 (0)
cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Data from the first 25 patients enrolled in this study was analyzed. However, recruitment was thought to be affected by the COVID-19 pandemic. The investigator intended to resume recruitment of the remainder of the sample, however additional funding was not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT04027049/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT04027049/ICF_001.pdf